CLINICAL TRIAL: NCT02399176
Title: Yoga in the Treatment of Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manhattan Physical Medicine and Rehabilitation, LLP (Other)
Collaborators: New York University (Other)
Responsible Party: Principal Investigator, Loren M. Fishman,MD, Loren M. Fishman, MD, Manhattan Physical Medicine and Rehabilitation, LLP
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2015-03-22; First posted 2015-03-26 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Yoga
MeSH Terms: conditions — Osteoporosis | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yoga of minimal intensity (Experimental): Does Yoga: At least 4 times/week.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — Subjects assume 10 physical postures for 30 seconds each
  Other Names: Iyengar Yoga

SUMMARY:
The study measures change in bone mineral density by the DEXA scan before and two or more years after beginning ten minutes of daily yoga designed to put pressure on the spine, hips and femur.

DETAILED DESCRIPTION:
After collecting blood and urine samples, and pre-study DEXA scans, qualifying patients are given an entry DEXA scan and a DVD with instructions to advance from beginner versions of 12 Iyengar-style yoga poses to more advanced levels in daily practice for 2 years. fter two years or more, subsequent DEXA scans are recorded. Interested participants are also encouraged to have hip and spine X-rays, and bone quality studies on study entry and two years later. Actual subject participation, intercurrent illnesses, fractures and changes in medication are self-monitored with an on line scorecard, supplemented by emails and/or telephone calls when judged necessary by the PI. Results are calculated by change in bone mineral density in the lumbar spine, hips and femurs by the DEXA scan, changes in osteoarthritis according to the X-rays, and changes in bone quality before and two or more years after beginning the ten minutes of daily yoga. Dose-response relationships between the amount and intensity of yoga practice and bone mineral density and quality are sought. Yoga-related fractures and other adverse effects are also noted.

ELIGIBILITY:
Inclusion Criteria:

* Past DEXA scan and, all within 6 months of study entry, DEXA scan and normal values for: Metabolic panel, TSH, PTH, ESR (or CRP), Vitamin D 25 hydroxy, Vitamin D 1,25 dihydroxy, Urine NTX.

Exclusion Criteria:

* Known metabolic bone disease such as osteogenesis imperfecta, current treatment with steroids, chemotherapy, or currently healing fractures of lumbar spine, hips or femurs.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 741 (Actual)
Dates: Start 2005-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
DEXA T-score | 2 years
  Bone mineral density change in spine, hip and femur after 2 years of yoga.

SECONDARY OUTCOMES:
Change in bone quality after doing yoga for two years. | two years
Number of fractures occurring while in study | two years

CONTACTS AND LOCATIONS:
Overall Officials: Loren M Fishman, MD, Principal Investigator — Manhattan Physical Medicine and Rehabilitation, LLP
Locations (1):
- Manhattan Physical Medicine and Rehabilitation, LLP, New York, New York, United States

REFERENCES:
- [Result] Fishman, LM. "Yoga for Osteoporosis - A pilot study." Topics in Geriatric Rehabilitation Vol. 25, No. 3, 2009 pp. 244-250.
- See also: Helpful site to learn more and to sign up for study. — http://sciatica.org